CLINICAL TRIAL: NCT03401970
Title: Dietary Carbohydrate and Internal Body Fat Mass in Women and Men With Obesity
Brief Title: Dietary Carbohydrate and Internal Body Fat
Acronym: CARBFUNC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/621
Record Dates: First submitted 2017-08-23; First posted 2018-01-17 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Adiposity
Keywords: Body composition; Internal body fat; Dietary pattern; Dietary carbohydrate
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acellular carbohydrate diet (Active Comparator): Prescribed dietary pattern. Carbohydrates from acellular sources, e.g., refined flour/bakery products, at least 500 grams of fruits/vegetables per day, and a macronutrient composition within typical nutritional recommendations for the general population.
  Interventions: Behavioral: Acellular carbohydrate diet
- Cellular carbohydrate diet (Experimental): Prescribed dietary pattern. Carbohydrates from cellular sources, e.g., root vegetables, fruits, whole-grain rice, non-flour grain products, at least 500 grams of fruits/vegetables per day, and a macronutrient composition within typical nutritional recommendations for the general population similar to the acellular carbohydrate diet.
  Interventions: Behavioral: Cellular carbohydrate diet
- Low-carbohydrate high-fat diet (Experimental): Prescribed dietary pattern. Energy largely from fat, cellular carbohydrate sources, and otherwise similar food types as in the acellular/cellular carbohydrate diets including at least 500 grams of fruits/vegetables per day.
  Interventions: Behavioral: Low-carbohydrate high-fat diet

INTERVENTIONS:
Behavioral: Acellular carbohydrate diet — Participants will be asked to consume 2,000 - 2,500 kcals, thereof 45 energy percent (E%) carbohydrate (up to 5 E% added sugar), 30 E% fat (10-12 E% saturated fatty acids and 7-10 E% polyunsaturated fatty acids) and 17 E% protein. They will use an original online/smartphone application that provides choices of meals/food combinations/recipes corresponding to their prescribed macronutrient profile and dietary pattern. Participants are asked to complete 3-day dietary records every 14 days throughout the study, and to report any deviations from the planned interventions.
  Arms: Acellular carbohydrate diet
Behavioral: Cellular carbohydrate diet — Participants will be asked to consume 2,000 - 2,500 kcals, thereof 45 energy percent (E%) carbohydrate (up to 1 E% added sugar), 38 E% fat (10-12 E% saturated fatty acids and 7-10 E% polyunsaturated fatty acids) and 17 E% protein. They will use an original online/smartphone application that provides choices of meals/food combinations/recipes corresponding to their prescribed macronutrient profile and dietary pattern. Participants are asked to complete 3-day dietary records every 14 days throughout the study, and to report any deviations from the planned interventions.
  Arms: Cellular carbohydrate diet
Behavioral: Low-carbohydrate high-fat diet — Participants will be asked to consume 2,000 - 2,500 kcals, thereof 10 energy percent (E%) carbohydrate (up to 1 E% added sugar), 73 E% fat (30 E% saturated fatty acids and 7-10 E% polyunsaturated fatty acids) and 17 E% protein. They will use an original online/smartphone application that provides choices of meals/food combinations/recipes corresponding to their prescribed macronutrient profile and dietary pattern. Participants are asked to complete 3-day dietary records every 14 days throughout the study, and to report any deviations from the planned interventions.
  Arms: Low-carbohydrate high-fat diet

SUMMARY:
This is a 2-year randomized controlled trial to test the effect of dietary carbohydrates, both quality and quantity, on changes in internal body fat mass. Up to 250 women and men with obesity are recruited in Bergen, Norway, and randomized to one of the following normo- and isocaloric dietary patterns (same amount of protein, polyunsaturated fatty acids and moderate energy, 2,000 - 2,500 kcal per day): 1) a low-fat high-carbohydrate diet primarily with refined (e.g., flour-based) carbohydrate sources, 2) a low-fat high-carbohydrate diet based on minimally refined (e.g., cellular) carbohydrate sources, and 3) a very-high-fat low-carbohydrate diet.

DETAILED DESCRIPTION:
Obesity, and high internal fat storage in particular, represents a tremendous and increasing health challenge across the world, and is linked to the recent introduction and globalization of an ultra-processed food supply largely based on refined carbohydrates. However, more high-quality studies are needed to directly assess the role of carbohydrate quality in abdominal adiposity. We also need studies with greater long-term adherence to prescribed food profiles, which may be achievied with the help of new electronic tools such as meal planning applications.

The participants select and plan all meals among a list of carefully designed options, using an application/recipe booklet developed for the study. Each recipe/meal/snack is designed to fully comply with the overall macronutrient- and dietary profile for the respective groups. We will further instruct the participants to record their meal choices during three days every 14 days, and to record all deviations throughout the intervention.

Enrolled participants are invited to study visits at baseline and after 3, 6, 9, 12 and 24 months. At all or some of these time points, the participants provide biological samples (blood, urine and feces, and for some, adipose and/or muscle tissue) and undergo phenotyping, e.g., measurement of body weight and fat mass by bioelectrical impedance analysis and low-radiation CT imaging, and a standardized meal test with blood sample collection up to 4 hours postprandially. In addition, participants will be asked to fill out a collection of questionnaires that assess quality of life, motivation, fatigue, gastrointestinal health, appetite and physical activity. We ask the participants to maintain the same level of physical activity throughout the study.

The primary outcome measure is change in internal body fat mass (visceral adipose tissue) measured by CT imaging. Secondary outcome measures include change in 2-hour postprandial serum concentrations of insulin, change in 4-hour postprandial serum concentrations of triacylglycerols, and change in fecal microbiota composition measured by 16S sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Body-mass index (BMI) equal to or above 30 kg/m2 and/or waist circumference equal to or above 102 cm for men and 88 cm for women
* Weight stable during the last 2 months before start of the study (less than 5 % change in body weight up or down)
* No known diabetes or consumption of diabetes medication
* Desire to follow a specified dietary pattern using specific recipes throughout the time of the study period
* Ability to periodically record food intake using a specially designed app for the study

Exclusion Criteria:

* Use of statins and/or diabetes medication
* Recent surgical or antibiotics treatment during the last 2 months before start of the study
* Chronic inflammatory bowel disease
* Serious disease
* Smoking
* Pregnancy or breast feeding
* Alcohol consumption during the study of more than 2 alcohol units per day (1 unit = 15 ml (12.8 g) pure alcohol)

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2021-03-24 (Actual)

PRIMARY OUTCOMES:
Change in internal body fat | Baseline and 6, 12 and 24 months
  Visceral fat mass (cm3) measured by computed tomography (CT) imaging

SECONDARY OUTCOMES:
Change in postprandial insulin | Baseline and 3, 6, 9, 12 and 24 months
  Circulating insulin concentrations measured before and 2 hours after intake of a standardized mixed meal
Change in postprandial C-peptide | Baseline and 3, 6, 9, 12 and 24 months
  Circulating C-peptide concentrations measured before and 2 hours after intake of a standardized mixed meal
Change in postprandial triacylglycerol | Baseline and 3, 6, 9, 12 and 24 months
  Triacylglycerol concentrations measured before and 4 hours after intake of a mixed meal
Change in postprandial area under the curve (AUC) glucose | Baseline and 3, 6, 9, 12 and 24 months
  Circulating glucose measured before and after 30, 60, 90, 120 and 240 minutes after intake of a standardized mixed meal
Change in postprandial non-esterified fatty acids | Baseline and 3, 6, 9, 12 and 24 months
  Circulating non-esterified fatty acid concentrations before and after 60, 120 and 240 minutes after intake of a standardized mixed meal
Change in fecal microbiome composition | Baseline and 3, 6, 9, 12 and 24 months
  Microbiome composition measured by 16S sequencing
Change in liver density | Baseline and 6, 12 and 24 months
  Calculated as liver/spleen attenuation index (Hounsfield units) based on quantification by computed tomography (CT) imaging
Change in pericardial fat mass | Baseline and 6, 12 and 24 months
  Pericardial fat mass (cm3) measured by computed tomography (CT) imaging
Change in abdominal subcutaneous fat mass | Baseline and 6, 12 and 24 months
  Abdominal subcutaneous fat mass (cm3) measured by computed tomography (CT) imaging
Change in coronary artery calcification (CAC) | Baseline and 6, 12 and 24 months
  CAC score calculated based on computed tomography (CT) imaging
Change in waist circumference | Baseline and 3, 6, 9, 12 and 24 months
  Waist circumference (cm) measured by a measuring tape
Change in body-mass index | Baseline and 3, 6, 9, 12 and 24 months
  Body-mass index measured as body weight (kg) divided by height (m) squared
Change in fasting insulin | Baseline and 3, 6, 9, 12 and 24 months
  Circulating fasting insulin concentrations
Change in fasting C-peptide | Baseline and 3, 6, 9, 12 and 24 months
  Circulating fasting C-peptide concentrations
Change in fasting TAG | Baseline and 3, 6, 9, 12 and 24 months
  Circulating fasting triacylglycerol concentrations
Change in fasting HDL cholesterol | Baseline and 3, 6, 9, 12 and 24 months
  Circulating fasting high-density lipoprotein cholesterol (HDL-C)
Change in TAG/HDL-C ratio | Baseline and 3, 6, 9, 12 and 24 months
  The ratio of circulating fasting triacylglycerol (TAG) and high-density lipoprotein cholesterol (HDL-C)
Change in fasting LDL cholesterol | Baseline and 3, 6, 9, 12 and 24 months
  Circulating fasting low-density lipoprotein cholesterol (LDL-C)
Change in apolipoprotein profile | Baseline and 3, 6, 9, 12 and 24 months
  Circulating fasting apolipoprotein profile measured by multiplex ELISA
Change in circulating and urine metabolites associated with one-carbon metabolism | Baseline and 3, 6, 9, 12 and 24 months
  Circulating metabolites in the serine, glycine and histidine pathways measured in the fasted state by GC-MS/MS
Change in total fat mass | Baseline and 3, 6, 9, 12 and 24 months
  Total fat mass measured by bioimpedance analysis (BIA)
Change in lean mass | Baseline and 3, 6, 9, 12 and 24 months
  Lean mass will be measured by bioimpedance analysis (BIA)
Change in appetite/fullness | Baseline and 3, 6, 9, 12 and 24 months
  Subjective appetite and fullness assessed and quantified by the VAS questionnaire
Change in gastrointestinal symptoms by the Roma III questionnaire | Baseline and 3, 6, 9, 12 and 24 months
  Gastrointestinal health will be surveyed and quantified by a questionnaire (Rome III Diagnostic Criteria for Irritable Bowel Syndrome (IBS)). The questionnaire surveys criteria for diagnosis of IBS within a 12-week period. The criteria for IBS are based on recurrent abdominal pain or discomfort, 3 days per month in the last 3 months (12 weeks), associated with ≥2 of the following criteria: 1.Improvement with defecation; 2. Onset associated with a change in stool frequency; 3. Onset associated with a change in stool form (appearance). The criteria are fulfilled with symptoms onset 6 months prior to diagnosis.
Change in gastrointestinal symptoms by the IBS-SSS questionnaire | Baseline and 3, 6, 9, 12 and 24 months
  Gastrointestinal health will be surveyed by the IBS-SSS questionnaire. Scores on the IBS-SSS range from 0 to 500 with higher scores indicating more severe symptoms. Subjects can be categorized as having mild (75-175), moderate (175-300), or severe (>300) IBS. A decrease of 50 points is associated with a clinically meaningful improvement. Each question on the VAS ranges from 0-100mm, where higher score indicates more severe symptoms.
  The categorization based on scores (total possible score = 500) are as follows:
  0-75 = not IBS 75-175= mild IBS 175-300 = moderate IBS 300-500 = severe IBS
Change in fatigue | Baseline and 3, 6, 9, 12 and 24 months
  The Fatigue Impact Scale will be used to compute a total score for fatigue by summing up the scores for subclasses as follows: cognitive functioning (10 items, subscale range: 0-40), physical functioning (10 items, subscale range: 0-40), and psychosocial functioning (20 items, subscale range: 0-80). The statements are ranged on a five-level scale (0 = no problem to 4 = extreme problems), giving a maximum total FIS score of 160 (total scale range: 0-160) where low scores indicate less fatigue-related issues.
Change in perception of health / quality of life | Baseline and 3, 6, 9, 12 and 24 months
  Obesity-specific quality of life is measured with "Patient-Reported Outcomes in Obesity" (PROS), which consists of 8 items tapping how different life domains are affected by obesity. PROS have one overall score, ranging from 0 (optimal) to 3 (poorest).
  Generic health-related quality of life is measured with RAND-36, which consists of dimensions ranging from 0 (poorest) to 100 (optimal). There are 8 subscales; physical functioning, physical role functioning, bodily pain, general health, vitality, social functioning, emotional role functioning and mental health. In addition, RAND-36 also have 2 summary scores: the physical component summary (PCS) (tapping from physical functioning, physical role functioning, bodily pain and general health) and mental component summary (MCS) (tapping from vitality, social functioning, emotional role functioning and mental health).
Change in quality of life related to gastrointestinal symptoms | Baseline and 3, 6, 9, 12 and 24 months
  The SF-NDI (Short-Form Nepean Dyspepsia Index (SF-NDI)) questionnaire will be used to assess quality of life / psychological wellbeing related to gastrointestinal symptoms. The 10-item SF-NDI was constructed and validated in patients with functional gastrointestinal disorders for measuring health-related quality of life. The 10-item short form includes five subscales: tension, interference with daily activities, eating/drinking, knowledge/control, and work/study, and each subscale contains two items. The items were measured by a 5-point graded Likert scale from 1 to 5. A total sum score for quality of life and a sum score for each of the five subscales were calculated by adding up scores for each item (range of total quality of life, 10-50; range of each subscale, 2-10). Higher scores indicate worse functioning or symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Simon N Dankel, PhD, Principal Investigator — University of Bergen; Gunnar Mellgren, MD PhD, Study Director — Haukeland University Hospital
Locations (1):
- Forskningsenhet for helseundersøkelser (research unit for clinical trials), Department of Clinical Science, University of Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jensen C, Sommersten CH, Laupsa-Borge J, Storas I, Valeur J, Mellgren G, Dierkes J, Dankel SN, Lied GA. Quality and quantity of carbohydrates, faecal short-chain fatty acids and gastrointestinal symptoms - results from a randomised, controlled trial (CARBFUNC). Clin Nutr. 2025 Jan;44:54-64. doi: 10.1016/j.clnu.2024.11.041. Epub 2024 Nov 26. PMID 39631208
- [Derived] Sommersten CH, Gjerde ES, Laupsa-Borge J, Andersen AI, Lawrence-Archer L, McCann A, Hansson P, Raza GS, Herzig KH, Lied GA, Martins C, Mellgren G, Dierkes J, Dankel SN. Relationship between Ketones, Ghrelin, and, Appetite on Isocaloric Diets with Varying Carbohydrate Quality and Amount: Results from a Randomized Controlled Trial in People with Obesity (CARBFUNC). J Nutr. 2023 Feb;153(2):459-469. doi: 10.1016/j.tjnut.2022.12.030. Epub 2022 Dec 29. PMID 36894239
- [Derived] Sommersten CH, Laupsa-Borge J, Andersen AIO, Fasmer KE, Holmefjord MA, Revheim I, Johannessen KK, Naesheim NT, Storas I, Leikanger T, Amundsen K, Skjerve KL, Lawrence-Archer L, Spjelkavik C, Haldorsen I, Lindseth I, Dierkes J, Mellgren G, Dankel SN. Diets differing in carbohydrate cellularity and amount similarly reduced visceral fat in people with obesity - a randomized controlled trial (CARBFUNC). Clin Nutr. 2022 Oct;41(10):2345-2355. doi: 10.1016/j.clnu.2022.08.028. Epub 2022 Sep 5. PMID 36116147